CLINICAL TRIAL: NCT04389905
Title: Equal Oral Health in Children: The Hageby-model
Acronym: EOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mats Bågesund (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Mats Bågesund, Associate Professor, PhD, Assistant Professor, Research Counselor, Senior Consultant Specialist in Pediatric Dentistry, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EquHag 2012; Dnr 2012/259-31 (Other: Regional Ethical Board Linköping); Dnr 2018/367-32 (Other: Regional Ethical Board Linköping)
Record Dates: First submitted 2020-04-24; First posted 2020-05-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries in Children; Economic Problems; Infant Conditions; Child, Preschool; Pregnancy Related; Educational Problems; Risk Reduction
Keywords: Dental Caries in Children; Pregnancy; Infant Conditions; Economic Problems; Child, Preschool; Health Education, Dental
MeSH Terms: conditions — Risk Reduction Behavior; Health Education | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized case control study following a cohort, of Children - whose mothers received extended oral health education from (before) birth until their 3-year dental examination - until their 6-year examniation, and comparing the results (e.g. caries experience and economical aspects) with a control group of age-matched individuals born during the same period.
  The study group of pregnant mothers (and their children) at the local Public Dental Clinic will be compared to a group of other pregnant mothers (and their children) and pregnant mothers (and their children) from the other dental clinics in the city and from another Public Dental Clinic with similar socioeconomic problems and similar caries prevalence as the clinic of the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Interviewing Oral Health Education Group (Experimental): The intervention group focused on the mothers from before birth until their child reached the age of 3 years. They received repeated questionnaires and repeated oral health education using the Motivational Interviewing (MI) technique.
  Interventions: Behavioral: Dental education - Motivational Interviewing
- Local Control Group (No Intervention): The local control group included other mothers and their children, who were (randomized according to) born during the same time as the children in the intervention group. They received only a questionnaire before their children were born. Caries data from 3- and 6-year examination is used.
- Similar Socio-economics Control Group (No Intervention): This control group is from a Public Dental Clinic with similar socioeconomics (among the families in the catchment area of the clinic) as in the intervention group. This control group included mothers and their children, who were (randomized according to) born during the same time as the children in the intervention group. They received only a questionnaire before their children were born. Caries data from 3- and 6-year examination is used.

INTERVENTIONS:
Behavioral: Dental education - Motivational Interviewing — Motivational Interviewing - Focusing on oral/dental health
  Other Names: Questionnaire
  Arms: Motivational Interviewing Oral Health Education Group

SUMMARY:
Pregnant women - living in thecatchment area of a public dental clinic with known higher caries experience and generally lower socioeconomical status than at other dental clinics in the Region - are recruited for the study.

Repeated information and surveys of dental knowledge, dental habits and medical conditions etc. is sample.

Before birth, one month after birth, and 12 and 18 months after birth of the Child, the mother repeatedly answers questionnaires and recieves information about dental care.

At 18 months,and at the 3- and 6-year dental examinations the caries experience dmft/deft is registered.

All Children and accompanying parent receives an individual caries preventive program between the examinations.

Evaluation will be focused on possible caries sreduction and Health econimic aspects of the interventions.

DETAILED DESCRIPTION:
1. At the first visit to maternal health care: Preliminary caries risk assessment of the family using questionnaire 1 to the expectant mother and father / partner. The invitation and time are given for an initial health call. The invitation is translated into the most common languages in Hageby and Navestad. If a translation into the current language is missing, an interpreter is hired.
2. During pregnancy: Health talk with specially trained dental hygienist / dental nurse at the local Public Dental Clinic (Folktandvården Hageby). Determination of the family's risk assessment in accordance with the criteria of the regional Public Dental Service in the County of Östergötland is adapted for the project.
3. One-month monitoring in child health care: Follow-up of caries risk assessment of the family with the help of questionnaire 2 to future mother and father / partner.
4. Care program 6-18 months with different designed depending on caries risk.
5. At 12 months: Group information or individual call, depending on risk, in collaboration with child health care. Follow-up of the family's caries risk assessment with questionnaire 3 to the expectant mother and father / partner.
6. At 18 months regardless of risk: Health talk, examination and renewed caries risk assessment of the child according to the criteria of the Public Dental Service.
7. Dental care program 18-30 months, individually designed depending on caries risk evaluation: Oral health behavior is evaluated using a caries risk assessment questionnaire. The questions in the form are based on factors that are of importance for caries development, and are supplemented with information from the maternity care and social services medical records. The questionnaire is constructed with yes and no as a response alternative, where the no-answers, together with an assessment of a dietary registration, indicate an increased risk of developing caries. The questionnaire registers risk behavior as a point. The evaluation is conducted as an assessment of changed risk points. The baseline data uses the score from the first questionnaire to be answered during pregnancy, according to point 1 above in the dental care program. The questionnaire is constructed based on known risk factors for caries, but has not been validated for measuring oral health behavior. A validation is therefore planned to be implemented as part of the project and applied for separately. Caries prevalence is evaluated by routinely collected caries epidemiological data when the children are 3 and 6 years and reported as the proportion of caries-free children, average dmft (= caries, extracted and filled teeth) and proportion of children with deft> =5. Three and six years are so-called indicator ages for caries epidemiological records. This means that caries data at the personal number level for all children in Östergötland are reported to the County Council. Participation in the dental care program is reported as the proportion of pregnant women who participate in the first health call compared to the proportion of pregnant women in control group 1 who participate in maternal health care's regular parental education on oral health at the midwifery. The usefulness of the questionnaire as a screening instrument is evaluated by comparing the outcome of the risk assessment with the caries outcome when the children in the control group are 3 and 6 years, respectively. The health economic evaluation focuses on cost efficiency. All costs associated with the intervention are recorded and calculated. Effects are calculated in the form of the number of people who come to the health interviews and meetings, changes in behavior, and in the longer term the changes in the number of dmft that occur. Cost efficiency is therefore calculated as the extra cost incurred per extra power (e.g. cost per person coming or cost per prevented dmft). The evaluation mainly uses a socio-economic perspective, which means that all costs and effects that arise at different levels in society are taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman visiting maternal health care at the Vrinevi Hospital, Norrköping, for the current pregnancy during the time of the study.
* The expecting mother's accommodation - during the time of the study - is at an address within Hageby and Navestad (defined as associated socio-economic cluster status 5). (Socio-economic affiliation).
* The participating Child must be examined in the Public Dental Service at the 3- and 6-year examinations.

Exclusion Criteria:

* Other home address than mentionned above.
* Moved out of the area during the time of the study.

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 667 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Early Childhood Caries (ECC) experience/prevalence at 3-years age | The outcome of ECC experience/prevalence is evaluated at 3-years age
  Early Childhood Caries experience/prevalence (dmft/deft)
Early Childhood Caries (ECC) experience/prevalence at 6-years age | The outcome of ECC experience/prevalence is evaluated at 6-years age
  Early Childhood Caries experience/prevalence (dmft/deft)

SECONDARY OUTCOMES:
Cost-benefit analysis of the intervention. | Evaluated when the child is 6 years old.
  Evaluate if the (private and public) cost for intervention (using MI Health education during the intervention from pregnancy until the child reaches the age of 3 years) are higher than the gain - measured as total (private and public) cost for each avoided dental treatment (e.g. filling or extraction) due to dental caries. The assessments will be based on Clinical assumptions of time and estimations of private cost.

OTHER OUTCOMES:
Change in Oral Health related knowledge level among mothers (after MI Health Education). | Baseline questionnaire answered before birth compared to [possible change in percentage correct answers] after 12 months
  Changed percentage of correct answers to questions in Questionnaire [Repeated use of a regionally designed questionnaire will be used to evaluate if the mothers' level of oral health related knowledge will change following the intervention.]

CONTACTS AND LOCATIONS:
Overall Officials: Mats Bågesund, Assoc Prof, Principal Investigator — Linköping University / Region Östergötland
Locations (1):
- Mats Bågesund, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No